CLINICAL TRIAL: NCT06466005
Title: UnityPhilly Response App for Overdose Reversal: Assessing Citywide Effectiveness and Sustainability
Brief Title: UnityPhilly Response App for Overdose Reversal
Status: Not yet recruiting | Type: Observational
Sponsor: Drexel University (Other)
Collaborators: University of Michigan (Other); Bar Ilan University (Unknown)
Responsible Party: Principal Investigator, Stephen Lankenau, Professor, Drexel University
Other Study IDs: 2401010340
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Active non-medical opioid user: Person who has used an opioid, e.g., heroin, fentanyl, non-medically in the past 30 days.
  Interventions: Other: UnityPhilly app
- Active prescription medical opioid user: Person who has used an opioid, e.g., hydrocodone, with a medical prescription in the past 30 days.
  Interventions: Other: UnityPhilly app
- Person in recovery from opioid misuse: Person who formerly used opioids non-medically and/or is on opioid replacement therapy.
  Interventions: Other: UnityPhilly app
- Caregiver/family members of groups 1, 2, 3: Person who is caring for or a family member of active non-medical user, medical user, or person in recovery.
  Interventions: Other: UnityPhilly app
- Concerned community member: Person in the community who is concerned about the opioid overdose crisis and is interested addressing the problem.
  Interventions: Other: UnityPhilly app

INTERVENTIONS:
Other: UnityPhilly app — UnityPhilly automatically connects bystanders and victims of opioid overdose with nearby community members who can respond immediately with naloxone.

SUMMARY:
The goal of this clinical trial is to discover if an overdose prevention app (UnityPhilly) can encourage citizen responders to respond and prevent opioid overdoses using the UnityPhilly app. The main hypotheses to answer are:

Hypothesis 1: UnityPhilly signal rates relative to EMS calls will increase over time. The primary outcome will be assessed as the total number of overdoses signaled by participants relative to all overdose-related EMS calls, per year.

Hypothesis 2: The number of cases where a nearby UnityPhilly participant successfully reverses an overdose with naloxone will increase over time. The primary outcome will be assessed as the number of successful reversals relative to the total number of responder arrivals, per year.

Participants will be supplied with the UnityPhilly app, training on how to use the app and respond to an opioid overdose using naloxone, and respond to follow up surveys about their experiences.

DETAILED DESCRIPTION:
This is a behavioral clinical trial, which is has been developed to evaluate and compare ways that people respond to a drug overdose using the UnityPhilly overdose response app. The UnityPhilly app, along with training participants how to use the app, the provision of naloxone, and overdose prevention training, is the intervention in this study. All individuals enrolled in this study are prospectively assigned to use the UnityPhilly app so that there is no control or placebo group - all receive the intervention. By enrolling five different types of individuals into the study, e.g., person who uses opioids, person in recovery, we will be evaluate the effectiveness of the UnityPhilly app in these different groups in responding to and reducing opioid overdose in Philadelphia. Aim 1 of the study will redevelop the UnityPhilly app previously tested in an earlier R34 study so that the app is easy to use among different groups of users in different overdose environments. Aim 2 of the study will enroll 450 study participants from 3 different neighborhoods in Philadelphia over a period of 9 months and who will be studied for an additional 12 month period to assess the effectiveness of the app. Participants will self-identify into the following 5 subgroups: (1) Active non-medical opioid user; (2) Active prescription medical opioid user; (3) Person in recovery from opioid misuse; (4) Caregiver/family member of (1), (2), or (3); or (5) Concerned community member. All 450 persons will be prospectively assigned to use of the UnityPhilly app into this longitudinal study. Effectiveness of the app, including such outcomes as overdoses signaled, willingness to respond to an app signal, and first to scene of an overdose, will be assessed among the five groups overtime using a mix of quantitative assessments (baseline, follow up, incident, log data) and qualitative interviews. Multivariate and qualitative analyses will assess a series of five hypotheses linked to key effectiveness outcomes. Aim 3 of the study will enroll an additional 3,000 resident volunteers to determine the sustainability of UnityPhilly using the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) Model. These 3,000 individuals, who will be exposed to the UnityPhilly app by the 450 study participants and/or other social media/community outreach during the study, will download/use the UnityPhilly app and will be assessed over a two-year period. Sustainability of the app, including reasons to join UnityPhilly, equity in diffusion of the app, network density of the app, will be assessed using a mix of quantitative assessments (baseline, log) and quantitative interviews from both the study participants (n=450) and resident volunteers (n=3,000). Multivariate and qualitative analyses (n=60) will assess a series of six research questions linked to key sustainability outcomes.

ELIGIBILITY:
Inclusion Criteria:

* owning a smartphone with a data package;
* living or working in one of three identified Philadelphia neighborhoods;
* aged 18 or older.

Exclusion Criteria:

* persons aged under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Key study enrollment criteria will include: owning a smartphone with a data package; living or working in one of three identified Philadelphia neighborhoods, i.e., Kensington, South Philadelphia, West Philadelphia; aged 18 or older. Furthermore, participants will be placed into one of the five subgroups based upon 30-day self-report of non-medical opioid use, medical opioid use, abstinence or recovery from any opioid use, family member or community self-affiliation (see subgroups 1-5 above). The study will enroll 450 participants and all will be assigned the intervention, i.e., UnityPhilly app.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Overdoses Signaled | 2 year period
  # events signaled by participants vs. # all overdose-related EMS calls, per year
Rate of Overdoses Reversed | 2 year period
  # successful opioid reversals vs. # all arrivals, per year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lankenau, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Even though the final datasets will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects based on advanced location analytics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Khalemsky M, Khalemsky A, Lankenau S, Ataiants J, Roth A, Marcu G, Schwartz DG. Predictive Dispatch of Volunteer First Responders: Algorithm Development and Validation. JMIR Mhealth Uhealth. 2023 Nov 28;11:e41551. doi: 10.2196/41551. PMID 38015602
- [Background] Ataiants J, Reed MK, Schwartz DG, Roth A, Marcu G, Lankenau SE. Decision-making by laypersons equipped with an emergency response smartphone app for opioid overdose. Int J Drug Policy. 2021 Sep;95:103250. doi: 10.1016/j.drugpo.2021.103250. Epub 2021 Apr 20. PMID 33887699
- [Background] Marcu G, Schwartz DG, Ataiants J, Roth A, Yahav I, Cocchiaro B, Khalemsky M, Lankenau S. Empowering communities with a smartphone-based response network for opioid overdoses. IEEE Pervasive Comput. 2020 Oct-Dec;19(4):42-47. doi: 10.1109/mprv.2020.3019947. Epub 2020 Nov 17. PMID 33568966
- [Background] Schwartz DG, Ataiants J, Roth A, Marcu G, Yahav I, Cocchiaro B, Khalemsky M, Lankenau S. Layperson reversal of opioid overdose supported by smartphone alert: A prospective observational cohort study. EClinicalMedicine. 2020 Aug 3;25:100474. doi: 10.1016/j.eclinm.2020.100474. eCollection 2020 Aug. PMID 32954238
- [Background] Marcu G, Aizen R, Roth AM, Lankenau S, Schwartz DG. Acceptability of smartphone applications for facilitating layperson naloxone administration during opioid overdoses. JAMIA Open. 2019 Dec 4;3(1):44-52. doi: 10.1093/jamiaopen/ooz068. eCollection 2020 Apr. PMID 32607487
- See also: UnityPhilly website — https://www.unityphilly.org/